CLINICAL TRIAL: NCT04889846
Title: Investigation of the Effectiveness of Family Collaborative Early Intervention Approach Based on Sensory Strategies, Activity Based Motor Training and Environmental Enrichment in Premature Infants: SAFE National Early Intervention Approach
Brief Title: The Effects of SAFE Early Intervention Approach in Premature Infants in Turkey
Acronym: SAFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Umut Apaydin, Research assistant, PhD, PT., Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-77082166-302.08.01-48434
Record Dates: First submitted 2021-05-09; First posted 2021-05-17 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Infant, Premature, Diseases
MeSH Terms: conditions — Infant, Premature, Diseases

STUDY DESIGN:
Intervention Model Description: Single blind randomised controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAFE early intervention group (Experimental): A family collaborative treatment program based on sensory strategies, activity-based motor training and environmental enrichment principles was created for the infants in the treatment group. Within the scope of the SAFE treatment approach, appropriate activities were explained to the families. Families were asked to do these activities every day for 10 weeks. The compliance of the families with the program was monitored every week via phone calls or the WhatsApp phone program. In addition, families were asked to keep a diary and note the duration of the activity. The homes of the families in the treatment group were visited at least once. During this visit, home environment was evaluated. In order to create an enriched home environment, families were informed about the toys and materials that can be obtained. The family's questions about the program were answered.
  Interventions: Procedure: SAFE early intervention approach
- Control group (Experimental): Within the scope of this study, the infants in the control group were given an NDT-based family training program in accordance with their corrected months and current functional levels. In this context, appropriate activities were taught to families. Families were asked to do these activities every day for 10 weeks. The compliance of the families with the program was monitored every week via phone calls or the WhatsApp phone program. In addition, families were asked to keep a diary and note the duration of the activity. One visit was made to the homes of the families in the control group. The family's questions about the program were answered.
  Interventions: Procedure: SAFE early intervention approach

INTERVENTIONS:
Procedure: SAFE early intervention approach — SAFE approach is a national early intervention approach which is based on sensory strategies, activity based motor training, family collaboration and environmental enrichment.

SUMMARY:
In this study, it was aimed to develop the SAFE treatment approach, which is a family collaborative early intervention approach based on sensory strategies, activity-based motor training and environmental enrichment, and to examine the effects of this approach on sensory, motor, cognitive and language development in premature infants.

DETAILED DESCRIPTION:
Early intervention practices in Turkey is widely based on the principle of neuro-developmental therapy (NDT). It has been reported in recent years that the NDT approach has minimal effect on the development of risky premature infants. For these reasons, it was necessary to develop an early intervention program that does not include passive interventions and includes sensory and motor strategies in our country.

Within the scope of this study, a new early intervention approach that can be applied to infants between 0-24 months has been developed based on the shortcomings in the literature. Sensory strategies, activity-based motor training, family collaboration and environmental enrichment constitute the basic principles of this early intervention program. The name of the early intervention program was formed from the English initials of these basic principles and was determined as SAFE early intervention approach (S: Sensory Strategies, A: Activity Based Motor Training, F: Family Collaboration, E: Environmental Enrichment).

In this study, it was planned to establish the theoretical and practical foundations of the SAFE early intervention approach developed by the Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation. Also we aimed to examine the effects of this approach on sensory, motor, cognitive and language development in preterm infants with corrected ages of 9-10 months.

ELIGIBILITY:
Inclusion Criteria:

* Being born before 37 weeks
* A history of Neonatal Intensive Care Unit (NICU) for 15 days or more
* Adjusted age to be between 9-10 months
* Family's willingness to participate in the study

Exclusion Criteria:

* Having a congenital anomaly or systemic disease
* Having a high risk for the diagnosis of Cerebral Palsy (Intraventriculer hemorrhage (IVH) Stage 4 or periventricular leukomalacia (PVL) Stage 3-4, such as the absence of fidgety movements).

Ages: 9 Months to 10 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-10-17 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
The Bayley Scales of Infant and Toddler Development, Third Edition (Bayley-III) | 10 weeks
  Bayley-III is a widely used test battery to assess cognitive, receptive and expressive language, gross and fine motor development in children aged 1 to 42 months. The items in each section are scored as 1 (can do the desired skill) and 0 (cannot do the desired skill). The raw scores obtained from all items are converted into scale points ranging from 1 to 19 points. Then, a composite score is obtained according to this scale score. It is the composite score commonly used in studies. Composite scores range from 40 to 160. The higher the score, the better the improvement.

SECONDARY OUTCOMES:
Hammersmith Infant Neurological Examination (HINE) | 10 weeks
  HINE is an easy-to-apply, standardized and scorable test used for clinical neurological evaluation of babies aged 2-24 months. The test consists of 3 parts. The first part is the scoring neurological examination section, which consists of 26 items that evaluate cranial nerve function, posture, movements, tone, reflexes and reactions. The second section is the motor milestones section and consists of 8 items that cannot be scored. The third part is the behavior section that cannot be scored and consists of 3 items. The first 26-item section can be scored as 0,1,2,3. The total score that can be obtained in HINE is 78. While the optimal score for 9-12 month infants is 73, this score is 70 for 6 month infants. Scores below 57 points per month indicate a great risk for the diagnosis of Cerebral Palsy (CP).
The Test of Sensory Functions in Infants (TSFI) | 10 weeks
  TSFI evaluates sensory processing and reactivity in infants aged 4-18 months. TSFI consists of 5 subtests: response to tactile deep pressure, adaptive motor response, visual-tactile integration, oculo-motor test, and response to vestibular stimulation. All subtests consist of a total of 24 items. The total score ranges from 0 to 49. In 10-12 month-old infants, a score between 44-49 indicates good sensory function, 41-43 points indicate risky status, 0-40 points indicate sensory processing problem.
Canadian Occupational Performance Measure (COPM) | 10 weeks
  Secondary outcomes included the COPM an individualised criterion-referenced measure of performance and satisfaction with performance of a parent-selected range of activities. In this study COPM was used at baseline to prioritise parent goals for their infants development and assess parents perception of their infants performance on identified goals and their own satisfaction with the infants current ability.
Affordances in the Home Environment for Motor Development - Infant Scale (AHEMD-IS) | 10 weeks
  Enrichment of the home environment was assessed with the AHEMD-IS. AHEMD-IS identifies opportunities available within the home to promote motor development, including characteristics of the indoor and outdoor environment and the presence of a range of toys and equipment. Total score possible for infants younger than 11 months is 66 while from 12 months possible total score is 93, to account for the expected increase in available learning materials.
The Depression, Anxiety and Stress Scales-Short Form (DASS-21) | 10 weeks
  DASS-21 is a questionnaire that evaluates the depression, anxiety and stress states of individuals. DASS-21 is a 21-item assessment tool developed from the 42-item long form of the scale. DASS-21 is specified as an easily applicable and low-cost scale. It has been shown to be effective in detecting patients with depressive and anxiety disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Bülent Elbasan, Prof, Study Director — Gazi University Faculty of Health Sciences
Locations (1):
- Gazi University Faculty of Health Sciences Department of Pyhsiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hielkema T, Blauw-Hospers CH, Dirks T, Drijver-Messelink M, Bos AF, Hadders-Algra M. Does physiotherapeutic intervention affect motor outcome in high-risk infants? An approach combining a randomized controlled trial and process evaluation. Dev Med Child Neurol. 2011 Mar;53(3):e8-15. doi: 10.1111/j.1469-8749.2010.03876.x. PMID 21291457
- [Background] Morgan C, Novak I, Badawi N. Enriched environments and motor outcomes in cerebral palsy: systematic review and meta-analysis. Pediatrics. 2013 Sep;132(3):e735-46. doi: 10.1542/peds.2012-3985. Epub 2013 Aug 19. PMID 23958771
- [Background] Morgan C, Novak I, Dale RC, Guzzetta A, Badawi N. Single blind randomised controlled trial of GAME (Goals - Activity - Motor Enrichment) in infants at high risk of cerebral palsy. Res Dev Disabil. 2016 Aug;55:256-67. doi: 10.1016/j.ridd.2016.04.005. Epub 2016 May 7. PMID 27164480
- [Background] Dusing SC, Burnsed JC, Brown SE, Harper AD, Hendricks-Munoz KD, Stevenson RD, Thacker LR, Molinini RM. Efficacy of Supporting Play Exploration and Early Development Intervention in the First Months of Life for Infants Born Very Preterm: 3-Arm Randomized Clinical Trial Protocol. Phys Ther. 2020 Aug 12;100(8):1343-1352. doi: 10.1093/ptj/pzaa077. PMID 32329778
- [Background] Pekcetin S, Aki E, Ustunyurt Z, Kayihan H. The Efficiency of Sensory Integration Interventions in Preterm Infants. Percept Mot Skills. 2016 Oct;123(2):411-23. doi: 10.1177/0031512516662895. Epub 2016 Aug 10. PMID 27511923